CLINICAL TRIAL: NCT01040182
Title: Polymorphism of Estrogen Genes in Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Hung-Yi Chiou, Ph.D./PI, National Science Council
Other Study IDs: NSC 97-2321-B-038-002
Record Dates: First submitted 2009-12-27; First posted 2009-12-29 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke patients
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Buffy coat and plasma will be retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ischemic stroke patients
- healthy subjects without cerebrovascular disease

SUMMARY:
The purpose of this study is to explore the association between the genetic polymorphisms of estrogen-related genes, including estrogen synthesis, metabolizing, and receptor genes, and ischemic stroke. Furthermore, independent and joint effects of traditional risk factors and estrogen related genes on risk of stroke in young adults will also be examined in this study.

DETAILED DESCRIPTION:
Cerebrovascular diseases are the third leading cause of death in Taiwan in 2007. It is also the most important reason for disability among elderly adults. Sex hormones are well reported to be associated with cardiovascular disease risk. Several studies showed that estrogens have been shown to have beneficial effects on the cardiovascular system via favorable effects on anti-inflammatory effects. Genetic polymorphisms of estrogen related genes are speculated to influence estrogen level and will count for human susceptible to risk of stroke in young adults. In addition, several studies showed that the decrease in estrogen-induced vascular inflammatory markers including adhesion molecules and chemokines might be the mechanism for vascular protection. Recently, a novel and unique mechanisms for 17β-Estradiol (E2) anti-inflammatory activity which is E2 prevents inflammatory gene transcription induced by inflammatory agents by inhibiting NF-κB intracellular transport was found. Therefore, we proposed a study to explore the association between the genetic polymorphisms of estrogen-related genes, including estrogen synthesis, metabolizing, receptor genes, and NF-κB and ischemic stroke in young adults.

ELIGIBILITY:
Inclusion Criteria:

* incident ischemic stroke patients diagnosed by CT or MRI.

Exclusion Criteria:

* non ischemic stroke patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 300 incident ischemic stroke patients will be recruited in the program project.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-11 (Estimated); Study Completion 2010-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Yi Chiou, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- WanFang Hospital, Taipei, Taiwan